CLINICAL TRIAL: NCT01672268
Title: Interest of Cardiac Computed Tomography (CT) to Optimize and Improve the Procedure of Transcatheter Aortic Valve Implantation (TAVI)
Brief Title: Interest of Cardiac Computed Tomography to Optimize and Improve the Procedure of TAVI
Acronym: CT-TAVI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-A001113-38; 2011-A001113-38 (Other: 2011-A001113-38)
Record Dates: First submitted 2012-04-18; First posted 2012-08-24 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2012-04

CONDITIONS: Aortic Stenosis
Keywords: cardiac computed tomography; Transcatheter Aortic Valve Implantation; safety and efficacy
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard TAVI procedure (Active Comparator): Patients without Cardiac CT measures before TAVI
  Interventions: Other: cardiac computed tomography
- Cardiac CT scan before TAVI procedure (Experimental): patients with cardiac CT measures before TAVI
  Interventions: Other: cardiac computed tomography

INTERVENTIONS:
Other: cardiac computed tomography — cardiac computed tomography, Transcatheter Aortic Valve Implantation, safety and efficacy
  Other Names: Transcatheter Aortic Valve Implantation

SUMMARY:
This is a pilot prospective, comparative, monocentric, randomized study with 2 groups. People with a severe aortic stenosis and a high risk of surgery are referred to a Trans catheter aortic valve implantation (TAVI).

DETAILED DESCRIPTION:
The proposed study is to show the interest of a cardiac computed tomography (CT) to improve the TAVI procedure. The Cardiac computed tomography (CT) shows the exact geometry of the aortic annulus and help the physician to find the right position of the prosthesis during the procedure. The hypothesis is that performing a cardiac CT before the TAVI could reduce the number of vascular peripheral complication, the number of stroke and can minimize the aortic regurgitation during the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a symptomatic severe aortic stenosis with a too high risk of surgical valvular replacement. This patient will be selected for a TAVI. In this study, we only randomized patient for a TAVI with an Edwards prosthesis
* male or female patient, older than eighteen years old
* who have given their written consent
* who are affiliated to the French social security system
* which has a too high risk of surgical valvular replacement (EuroSCORE logistic > 20% or Society of Thoracic Surgeons Score > 10, or contre indicated to a cardiac surgery by a heart team
* Severe Aortic stenosis with symptoms like dyspnea, heartache, syncope, heart failure

Exclusion Criteria:

* Patient who can't give his written consent because of his physical or mental status
* Adult patient protect by law (article L1121-8),
* Person deprived of liberty (article L1121-8),
* Pregnant women
* Patient in terminal phase of illness,
* Terminal kidney failure
* Allergy to iodine
* bicuspids ou unicuspid aortic,
* Diameter of the left ventricular outflow tract < 18mm or > 25mm,
* Diameter of the femoral artery < 7mm, tortuosity or calcifications
* Septal hypertrophy
* Apical thrombosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Composite end point | participants will be followed for the duration of 1 year
  Composite end point with Stroke (symptoms and CT or MRI), Vascular complications (hematoma with the need of transfusion, dissection of artery/ legs ischemia), and Aortic regurgitation after the procedure, evaluated by transthoracic echocardiography

SECONDARY OUTCOMES:
To compare results of transthoracic / transoesophageal echocardiography and cardiac CT | inclusion visit
  • Size of the aortic annulus/ diameter and area
To compare results of transthoracic / transoesophageal echocardiography and cardiac CT | inclusion visit
  • Left ventricular outflow tract, anatomy of the aortic roots
To compare results of transthoracic / transoesophageal echocardiography and cardiac CT | inclusion visit
  • Left ventricular function, size, volume

CONTACTS AND LOCATIONS:
Overall Officials: Gilles MD BARONE ROCHETTE, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France